CLINICAL TRIAL: NCT02321605
Title: Efficacy of Best Possible Self Intervention Over Time: A Randomized Control Trial
Brief Title: Efficacy of Best Possible Self Intervention Over Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaimeI08
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Best Possible Self Intervention
Keywords: Best Possible Self; Positive Psychology; Optimism; Positive Technology; Future Thinking
MeSH Terms: interventions — Activities of Daily Living

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BPS exercise (Experimental): Intervention group which requires people to envision themselves in a future in which all has gone in the best possible way.
  Interventions: Behavioral: e-BPS
- Daily Activities (Placebo Comparator): Control group which consists of thinking and writing about all the activities and situations that had taken place during the last 24 h.
  Interventions: Behavioral: Daily Activities

INTERVENTIONS:
Behavioral: e-BPS — Participants are asked to write and imagine about a future in which they have reached all their goals and they have developed all their potentialities in four different domains: personal, professional, social and health domain.
  They carry out the exercise in a Positive Technology System called the "Book of Life", which has shown efficacy in the enhancement of positive mood (Baños, Etchemendy, Farfallini, García-Palacios, Quero & Botella, 2014). This application looks like a personal diary, where participants can write all that they want and these essays are supported by multimedia content (pictures, songs and videos). Additionally, they can continue doing the exercise in a web platform in which they can visualize all the content they had developed previously.
  Other Names: Best Possible Self; Positive Psychology Intervention
  Arms: BPS exercise
Behavioral: Daily Activities — Participants are asked to think and write about all that they have done the last 24 hours. They carry out the exercise in a powerpoint document, where they can record all the activities, situations and thoughts.
  Other Names: Best Possible Self; Positive Psychology Intervention
  Arms: Daily Activities

SUMMARY:
This study is aimed to test the efficacy of a Positive Psychology Intervention (Best Possible Self) over optimism, future expectancies and positive affect at mid-term, in comparison to a control group. The principal hypothesis is that Best Possible Self intervention will enhance significantly the levels of optimism and positive affect in comparison to the control group at short and mid-term.

DETAILED DESCRIPTION:
Over the last fifteen years, research in the field of positive psychology has increased exponentially (Bolier, Haverman, Westerhof, Riper, Smit & Bohlmeijer, 2013; Sin & Lyubomirsky, 2009). These studies have shown that positive moods and positive emotions lead people to think, feel, and act in favor of their approach goals, promoting their involvement in them (Lyubomirsky, 2001). One of the main arms of this framework, is the development of exercises and treatment protocols aimed to promote the appearance of different positive emotions and states, called Positive Psychology Interventions (PPIs).

In this sense, Best Possible Self (BPS) has been included as a PPI, since is aimed to enhance wellbeing. Specifically, BPS is a positive future thinking technique, which requires people to envision themselves in the future, after everything has gone as good as it possibly could. This exercise has shown efficacy improving optimism, future expectancies and positive affect compared to a control condition, in general population (Meevissen, Peters & Alberts, 2011; Sheldon &Lyubomirsky, 2012; Peters, Flink, Boersma & Linton, 2010).

Furthermore, the progress of Information and Communication Technologies (ICTs), has allowed the development of technology applications and devices that could enhance the quality of experience and the wellbeing levels. This approach is called Positive Technology (PT) and it can be used as a complement to PPIs. PT can be defined as the scientific and applied approach to improve the quality of our personal experience trying to increase wellness and generate strengths (Riva, Baños, Botella, Wiederhold & Gaggioli, 2012).

Taking into account the prior literature, the aim of the present study is to carry out a randomized controlled study in order to replicate the findings about the effects of BPS on optimism, mood and affect in young general population. The exercise will be applied through a Positive Technology system and the effects will be analyzed during four months. The design employed in this study is similar to the used in other studies (Meevissen et al, 2011; Renner, Schwarz, Peters & Huibers, 2014; Sheldon & Lyubomirsky, 2006).

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 70 years old.
* Be willing to participate in the study.
* Have an e-mail address.

Exclusion Criteria:

* Presence of severe physical illness.
* Presence of psychological disorders.
* Be receiving psychological treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Subjective Probability Task (SPT; MacLeod, 1996). | 4 months
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 y 0.91, respectively).

SECONDARY OUTCOMES:
Positive and Negative Affect Scale (PANAS, Watson, Clark & Tellegen, 1988; Sandín et al., 1999). | 4 months
  This measure analyzes the levels of positive (PA) and negative affect (NA). The instrument consists of 20 items, 10 for each level of affect. Participants rate on a 5-point scale (Not at all - Extremely). The Spanish version has demonstrated high internal consistency (0.89 to 0.91 for PA and NA in women and 0.87 for AP and 0.89 for AN in men) in college students.
Life Orientation Test (Lot-R; Otero, Luengo, Romero Gómez & Castro, 1998; Scheier, Carver & Bridges, 1994). | 4 months
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 y 0.91, respectively).
Beck Depression Inventory II (BDI-II; Beck, 1996) | 4 months
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and test-retest reliability of around 0.8. The Spanish version of this instrument has also shown a high internal consistency (Cronbach's alpha of 0.87) for both the general and the clinical population (Cronbach's alpha of 0.89). Summed to obtain the total score, which can be a maximum of 63 points.

OTHER OUTCOMES:
Eysenck Personality Questionnaire - Revised - Neuroticism (EPQ-R-N; Eysenck, Eysenck & Barrett, 1985; Eysenck & Eysenck, 1997). | Baseline
  This scale assesses the neuroticism level of the individual, showing if he is stable or neurotic. This subscale is composed by 12 items of dicotomic response (yes-not). Regarding psychometric properties, Eysenck and Eysenck (1997) got an alpha coefficient between 0-73 and 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, Professor, Study Director — Universitat Jaume I; Juana M Bretón, Assistant Professor, Study Director — Universitat Jaume I; Angel Enrique, PhD student, Study Chair — Universitat Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

REFERENCES:
- [Background] Botella C, Riva G, Gaggioli A, Wiederhold BK, Alcaniz M, Banos RM. The present and future of positive technologies. Cyberpsychol Behav Soc Netw. 2012 Feb;15(2):78-84. doi: 10.1089/cyber.2011.0140. Epub 2011 Dec 9. PMID 22149078
- [Background] Meevissen YM, Peters ML, Alberts HJ. Become more optimistic by imagining a best possible self: effects of a two week intervention. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):371-8. doi: 10.1016/j.jbtep.2011.02.012. Epub 2011 Mar 2. PMID 21450262
- [Background] Peters, M. L., Flink, I. K., Boersma, K. y Linton, S. J. (2010). Manipulating optimism: Can imagining a best possible self be used to increase positive future expectancies? The Journal of Positive Psychology, 5(3), 204-211.
- [Background] Sheldon, K. M., y Lyubomirsky, S. (2006). How to increase and sustain positive emotion: The effects of expressing gratitude and visualizing best possible selves. The Journal of Positive Psychology, 1(2), 73-82.
- [Background] Baños, R. M., Etchemendy, E., Farfallini, L., García-Palacios, A., Quero, S., & Botella, C. (2014). EARTH of Well-Being System: A pilot study of an Information and Communication Technology-based positive psychology intervention. The Journal of Positive Psychology, 9(6), 482-488.
- See also: Laboratory of Psychology and Technology of the Universitat Jaume I — http://www.labpsitec.uji.es